CLINICAL TRIAL: NCT05617196
Title: Feasibility of a Virtually Delivered Preoperative Rehabilitation Program for Patients Awaiting TAVI to Reduce Frailty: The Virtual PREHAB Study
Brief Title: Virtual PREHAB Study for Patients Undergoing TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS-NHIG-2021-1905
Record Dates: First submitted 2022-10-26; First posted 2022-11-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases in Old Age; Frailty; TAVI
Keywords: Frailty; Virtual PREHAB; Cardiac rehabilitation; TAVI
MeSH Terms: conditions — Frailty | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator)
  Interventions: Behavioral: Standard care
- Virtual PREHAB (Experimental): In addition to standard care, participants randomized to the The virtual PREHAB program will be delivered by the Hearts and Health in Motion cardiac rehabilitation CR health care team including a medical director nurse, dietician, and physiotherapist who routinely deliver CR postoperatively. The virtual PREHAB program will be up to 8-weeks in duration and deliver the core components of CR online or by telephone.
  Interventions: Behavioral: Virtual PREHAB

INTERVENTIONS:
Behavioral: Virtual PREHAB — The Virtual PREHAB program begins with a virtual health care team assessment. The physiotherapist will support patients in identifying ways to safely engage in home-based physical activities and in their neighborhoods. Additional weekly 30-minute telephone consultations with the physiotherapist, nurse, and dietitian are provided as well as three 30-minute online consultations are provided; telephone calls will replace these online consults if the patient does not have internet access. Telephone and/or online consults with participants will monitor the progression of the individual through the program, review patient materials, review medication changes, as well as provide recommendations to adopting a physically active lifestyle, diet, well-being, smoking, or other supports available to the patient. Medication changes are monitored by a nurse and any necessary medication recommendations involve the program's medical director, the patient's family physician, and TAVI team.
  Arms: Virtual PREHAB
Behavioral: Standard care — In Nova Scotia, patients are referred to the TAVI program. The TAVI health care team, consisting of a cardiac surgeon, cardiologist, nurse, and geriatric team conduct patient assessments and provide guidance and resources on self management.Once patient assessments are completed, patients are discussed at a multidisciplinary team meeting. When a patient is accepted for TAVI, they are placed on a waiting list which lasts for 3-6 months depending on urgency.
  Arms: Standard Care

SUMMARY:
Nova Scotians are aging and many are becoming frailer. People with frailty are more likely to live in worse health and do not recover well from major events, such as open heart surgery. Many people are also too frail to receive open heart surgery. Less invasive procedures called transcatheter aortic valve implantation, or TAVI, are provided for the frailest patients. While TAVI is life-saving, frailer patients are less likely to survive in better health after their operation. Patients in Nova Scotia can also wait up to 3-6 months for their operation where they become frailer or can die before receiving TAVI. The investigators believe that it is important to support these individuals to improve their frailty and overall health before their operation.

Center-based cardiac rehabilitation is offered to patients after, but not before TAVI to improve their health. Center-based preoperative cardiac rehabilitation (i.e., PREHAB) can safely improve the function of frail patients who received open heart surgery. However, many patients cannot come to a center-based PREHAB because of transportation requirements to access the program. Another option is to support these patients with virtually delivered PREHAB, where they can stay in their homes. However, this possibility has not been studied.

For this study, virtual PREHAB will be delivered using the virtual cardiac rehabilitation program in Nova Scotia to patients before TAVI. This intervention will be delivered by healthcare providers who routinely care for TAVI patients, including a medical director, program lead, nurse, physiotherapist, and dietician. Ther goal of this study is to determine if it is feasible and safe to use virtual PREHAB to reduce frailty before TAVI. This research fits with Research Nova Scotia's priorities to improve patient outcomes in those with significant long-term health conditions, and to provide accessible, safe, and quality virtual healthcare to patients so they can thrive after their operation.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients attending the TAVI clinic at the Queen Elizabeth II Health Sciences Centre
* Informed written or verbal consent

Exclusion Criteria:

* New York Heart Association or Canadian Cardiovascular Score of 4
* Severe functional limitations
* Cognitive impairment that impacts consenting ability
* Significant language barrier
* No internet or telephone access that precludes virtual PREHAB participation

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CLSA-FI | Baseline
  Canadian Longitudinal Study on Aging Frailty Index; range 0-1 (lower is better)
CLSA-FI | 8-weeks preoperatively
  Canadian Longitudinal Study on Aging Frailty Index; range 0-1 (lower is better)
CLSA-FI | 1-week preoperatively
  Canadian Longitudinal Study on Aging Frailty Index; range 0-1 (lower is better)
CLSA-FI | 3-months postoperatively
  Canadian Longitudinal Study on Aging Frailty Index; range 0-1 (lower is better)
PFFS-FI | Baseline
  Pictorial-Fit Frail Scale Frailty Index; range 0-1 (lower is better)
PFFS-FI | 1-week preoperatively
  Pictorial-Fit Frail Scale Frailty Index; range 0-1 (lower is better)
PFFS-FI | 8-weeks preoperatively
  Pictorial-Fit Frail Scale Frailty Index; range 0-1 (lower is better)
PFFS-FI | 3-months postoperatively
  Pictorial-Fit Frail Scale Frailty Index; range 0-1 (lower is better)

SECONDARY OUTCOMES:
EQ-5D-5L health-related quality of life | Baseline
  Euroqol-5 dimension-5 level health-related quality of life; range 5-25 (lower is better)
EQ-5D-5L health-related quality of life | 8-weeks preoperatively
  Euroqol-5 dimension-5 level health-related quality of life; range 5-25 (lower is better)
EQ-5D-5L health-related quality of life | 1-week preoperatively
  Euroqol-5 dimension-5 level health-related quality of life; range 5-25 (lower is better)
EQ-5D-5L health-related quality of life | 3-months postoperatively
  Euroqol-5 dimension-5 level health-related quality of life; range 5-25 (lower is better)
VARC-3 Composite clinical end-points | Hospital discharge (assessed up to day 14)
  Valvular Academic Research Consortium V.3.0 clinical endpoints (Mortality, Neurologic events, Hospitalization, Rehospitalization, Bleeding and transfusions, Vascular and access-related complications, Cardiac structural complications, Other procedural or valve-related complications, New conduction disturbances and arrhythmias, New conduction disturbances and arrhythmias, Myocardial infarction, Bioprosthetic valve dysfunction, Leaflet thickening and reduced motion, Clinically significant valve thrombosis, Patient-reported outcomes and health status. Fewer complications indicate a better surgical outcome
VARC-3 Composite clinical end-points | 30-days postoperatively
  Valvular Academic Research Consortium V.3.0 clinical endpoints (Mortality, Neurologic events, Hospitalization, Rehospitalization, Bleeding and transfusions, Vascular and access-related complications, Cardiac structural complications, Other procedural or valve-related complications, New conduction disturbances and arrhythmias, New conduction disturbances and arrhythmias, Myocardial infarction, Bioprosthetic valve dysfunction, Leaflet thickening and reduced motion, Clinically significant valve thrombosis, Patient-reported outcomes and health status. Fewer complications indicate a better surgical outcome
Cardiac rehabilitation attendance | 3-months postoperatively
  Percent of people attending cardiac rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No